CLINICAL TRIAL: NCT04789759
Title: Comparative Clinical Performance of Biphasic Calcium Sulfate Cement Matrix With Hydroxyapatite Granules in a Socket Preservation Model: a Pilot Clinical Trial Parallel Group Assignment
Brief Title: Biomaterial Clinical Performance in a Socket Preservation Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Advanced Dentistry, Lisbon (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2021-02-13; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Bone Loss; Alveolar Bone Resorption
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: Case Series of 10 consecutive cases , with one extraction (at least ) with a type 2 socket, Control group, 10 consecutive dental extractions.
Who Masked: Outcomes Assessor
Masking Description: Person who does the volumetric analysis is blinded, Person who makes data treatment is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Socket Preservation Alloplastic Material (Experimental): 10 Consecutive Patients with hopeless teeth and 1/3 or more buccal bone resorption will be placed in a therapy go bone regeneration called socket preservation technique.
  The surgery will include placement of 2/3 biphasic calcium sulfate cement matrix's with hydroxyapatite (HA granules) to fill the alveolar defects, and place a resorbable membrane sutured to adjacent tissue, to avoid material leakage.
  No flap retraction. 3 Month later an implant will be placed, and a bone biopsy of the healed socket harvested. 2 Month later a final Zirconia ceramic crown screw retained to the osseointegrated implant.
  Primary (T0) and Secondary (T1) stability measured with ISQ values.
  Intraoral Scanner and an STL File will be taken at T0 , T1 and T2 for volumetric alteration evaluation.
  Interventions: Device: Socket Preservation - Bond Apatite synthetic bone substitute
- Extraction Socket Spontaneous Healing (Active Comparator): 10 Consecutive patients with a tooth extraction without the aim of placing a future implant and without Biomaterial filler placed in the socket. Spontaneous healing
  Interventions: Procedure: Socket healing - No Filler

INTERVENTIONS:
Device: Socket Preservation - Bond Apatite synthetic bone substitute — Pre-op CBCT scanner for evaluating bone conditions around hopeless tooth. If 1/3 of the buccal plate is missing, considered a class 2 alveolar socket.
  Extraction of tooth and place 2/3 biphasic calcium sulfate cement matrix's with Hydroxyapatite (HA granules) , condensed , and covered with a resorbable membrane suture to the adjacent tissue.
  At implant placement ,take bone for histological preparation and histomorphometric analysis of the healing pattern.
  At T0, T1 and T2 measure adjacent teeth periodontal status , Probing Depth , bleeding on probing.
  Volumetric measurements, will use fixed landmarks (ex. adjacent teeth) to calibrate the STL measurements. Calculate the difference between pre-extraction socket and the post treatment with the alloplastic material.
  Primary and secondary stability will be measured by ISQ units with a RFA machine, that will include the machine to measure and the magnetic tip to be screwed in the implant platform.
  Other Names: alveolar regeneration; bone regeneration
  Arms: Socket Preservation Alloplastic Material
Procedure: Socket healing - No Filler — Pre-op CBCT scanner for evaluating bone conditions around hopeless tooth, at extraction day, no flap opening , atraumatic extraction, no biomaterial filler, At T0, T2 measure adjacent teeth periodontal status , Probing Depth , bleeding on probing.
  Volumetric measurements will include an intramural scanner from all the stages , we will use fixed landmarks (ex. adjacent teeth) to calibrate the STL measurements. Calculate the difference between pre-extraction socket and the post treatment with the alloplastic material.
  Other Names: Alveolar Socket spontaneous healing
  Arms: Extraction Socket Spontaneous Healing

SUMMARY:
When a dental extraction is performed, sequential cascade of events happens that lead to a modeling and remodeling of the area.

This phenomenon leads to bone resorption and consequential volume loss atrophy. In literature several biomaterials (Autogenous, alloplastic, allografts and xenografts) were tested as alveolar fillers with the aim of controlling this physiologic event.

Socket preservation is today a very widely spread dental technic to preserve the alveolar dimensions, that uses a wide range of biomaterials.

Alloplastic materials have a fair evidence to work in several regenerative procedures in the oral and maxillofacial region.

This pilot trial aims to characterize Histologic bone healing pattern in a human socket preservation model of 2/3 biphasic calcium sulfate cement matrix's and Hydroxyapatite (HA granules).

Alterations in Volumetric alveolar socket changes in a socket preservation clinical model will also be studied.

DETAILED DESCRIPTION:
Aim : To evaluate histologic performance and volumetric outcome of a bone substitute used in dentistry for guided bone regeneration procedures.

Model : Human Socket preservation surgery with a control group of spontaneous alveolar healing.

Inclusion criteria includes a class 2 or 3 (loss of at least 1/3 of the buccal bone of the alveolar socket) post-extraction sockets.

Clinical Experimental Methodology :

Atraumatic extraction of the hopeless tooth without flap retraction, after socket mechanical debridement , fill with 2/3 biphasic calcium sulfate cement matrix's with Hydroxyapatite (HA granules) and covered with a resorbable membrane.

3 Month after a CBCT is performed for implant planning.

At implant placement a 2 mm trephine will be used for core extraction.

Measurements (Stl File) on the day of surgery (Baseline T0) and at implant placement (3 month after tooth extraction) (T1) and after delivery final crown (T2).

Discrepancy (Trueness) Between STL Files in Teeth Adjacent to Implant will be used at T0, T1 and T2.

Histologic measure comprise percentage of vital bone formation, fibrous/connective tissue, and material remnant, in a socket preservation model

To Measure Volumetric changes reverse engineering software (Geomagic Control X, 3D Systems) will be used.

Other evaluation parameters involve radiographic Cone Beam Computer Tomography evaluation, primary stability, implant survival and implant success rate

Clinical Control Methodology :

Atraumatic extraction of the hopeless tooth without flap retraction, after socket mechanical debridement Measurements (Stl File) on the day of surgery (Baseline T0) and at 3 month after tooth extraction) (T1) Discrepancy (Trueness) Between Standard Tessellation Language Files in Teeth Adjacent to Implant will be used at T0 and T1

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. requiring extraction of teeth in the premolar region and anterior maxilla (15-25), presence of intact 2/3 or less, buccal bone plate
3. ASA (Physical Status Classification System, American Society of Anesthesiologist) I or II.

Exclusion Criteria:

1. patients with uncompensated systemic diseases, metabolic and healing disorders, i.e. diabetes mellitus, hyperparathyroidism, cancer, HIV,
2. heavy smokers (>5 cigarettes/ day),
3. bone metabolic diseases,
4. severe renal dysfunction or liver disease,
5. had received systemic corticosteroids or other immunosuppressive agents, radiation therapy and/or chemotherapy for the past 2 months,
6. active infections in the surgical site
7. patients with periodontal or/and endodontic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Histologic Examination Histomorphometric Analysis | 3 month after tooth extraction
  Histologic measure, percentage of Vital Bone formation, Fibrous/connective tissue, and material remnant present in the sample.

SECONDARY OUTCOMES:
Volumetric Changes Clinical | at pre-extraction and at final crown insertion up to 1 year
  Measure Linear changes reverse engineering software (Geomagic Control X, 3D Systems) in mm.
Radiographic CBCT - Bone evaluation | at pre-extraction and at final crown insertion up to 1 year
  Measure Linear changes in bone from T0 baseline to Implant Placement T1 in mm
Primary and Secondary stability | at implant placement and at dental crown insertion up to 1 year
  Measure the Resonance Frequency Analysis at implants placed in regenerated bone
Incidence of Implant Success rate | at final treatment (crown insertion) up to 1 year
  Measure implant status peri-implant parameters , bleeding on probing in percentage of sites
Implant probing depth | At implant insertion and At final treatment (crown insertion) up to 1 year
  Measure the attachment loss in mm
Implant marginal bone loss. | at implant placement and at final crown insertion (up to 1 year)
  Measure bone position regarding Implant Platform
Incidence of Survival rate | at dental crown placement (final treatment) up to 1 year
  if the implant is osseointegrated

CONTACTS AND LOCATIONS:
Overall Officials: Andre Chen, Phd, Principal Investigator — International Advanced Dentistry; João Borges, Msc, Study Director — International Advanced Dentistry; Elena Cervino, Msc, Study Chair — International Advanced Dentistry; Amos Yahav, DMD, Study Chair — Augma Bio; Ofir Yahav, DMD, Study Chair — Augma Bio